CLINICAL TRIAL: NCT02434081
Title: A Phase II Trial Evaluating the Safety and Efficacy of the Addition of Concurrent Anti-PD 1 Nivolumab to Standard First-line Chemotherapy and Radiotherapy in Locally Advanced Stage IIIA/B Non-Small Cell Lung Carcinoma
Brief Title: NIvolumab COmbination With Standard First-line Chemotherapy and Radiotherapy in Locally Advanced Stage IIIA/B Non-Small Cell Lung Carcinoma
Acronym: NICOLAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: Bristol-Myers Squibb (Industry); Frontier Science Foundation, Hellas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETOP 6-14 NICOLAS; 2014-005097-11 (EudraCT Number); SNCTP000001672 (Registry Identifier: Swiss National Clinical Trials Portal (SNCTP))
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Results first posted 2021-10-25 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Non-small Cell Lung Cancer Stage III
Keywords: NSCLC; IIIA/B
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemo-radiotherapy with concurrent nivolumab (Experimental): 4 doses of nivolumab 360mg concurrently with standard chemo-radiotherapy, followed by 480mg for up to 1 year from start of nivolumab treatment.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is a fully human monoclonal antibody that targets the programmed death-1 (PD-1) cell surface membrane receptor. PD-1 is a negative regulatory molecule expressed by activated T and B lymphocytes.Binding of PD-1 to its ligands, 1 (PD-L1) and 2 (PD-L2), results in the down-regulation of lymphocyte activation. Nivolumab inhibits the interaction of programmed cell death Protein 1 (PD-1)with its ligands, PD-L1 and PD-L2, resulting in enhanced T-cell proliferation.
  Other Names: BMS-936558

SUMMARY:
The aim of the study is to investigate the tolerability (how severe the side effects are) and the efficacy (how well the treatment works) when nivolumab is added to the current standard treatment (chemotherapy and radiotherapy) given to patients with advanced NSCLC.

DETAILED DESCRIPTION:
Over the past decade, concomitant chemotherapy and radiotherapy has become the first choice treatment for most patients with stage III non-small-cell lung carcinoma (NSCLC).

However, only about 30% of patients are alive 5 years after con¬comitant therapy. These figures remain approximately the same with the addition of surgery. After chemo-radiotherapy, at least 30-40% of the patients show local tumour progression on CT scans as first site of relapse. Also after surgery, about 30% of patients fail locally as a first site of recurrence. In addition, more than half of the patients eventually develop distant metastases that may have been present but undetected at the time of staging or that may have come from persistent or recurring local disease. It is thus obvious that new approaches that preferentially tackle both local and distant disease sites are needed to improve long-term survival and cure rates.

Attempts to improve the long-term survival include radiotherapy dose escalation/acceleration, new chemotherapy combinations, and adding biological agents and cancer vaccines to standard regimens. At present, none of these have demonstrated an improved outcome.

Improved understanding of the immune profile of NSCLC has led to immunotherapeutic strategies, including inhibitory molecules responsible for abrogating an anti-cancer immune response such as PD-1 and CTLA-4. Nivolumab, an investigational monoclonal antibody that inhibits the immune checkpoint receptor PD-1 expressed on activated T cells, has demonstrated positive results in several trials in previously treated patients with advanced NSCLC. However, rare cases of severe or fatal pneumonitis have been reported throughout clinical trials using anti-PD1 or anti-PDL1 compounds.

Pre-clinical data consistently show a clear beneficial effect by combining local radiotherapy and anti-PD-1. Not only was the local tumour control increased, but an "abscopal" effect on distant metastases could be observed. Radiotherapy clearly acted as an "in situ" tumour vaccination resulting in the induction of specific anti-tumour immunity in all sites of the body that could result in a clinical anti-tumour effect because of the combination with anti-PD-1.

In these models, the concurrent administration of anti-PD-1/PD-L1 antibodies was more efficient to provoke an anti-tumour immune response than the sequential approach.

While the role of immunotherapy is currently being evaluated as monotherapy or in combination with chemotherapy or tyrosine kinase inhibitors in all lines of treatment of advanced NSCLC, as monotherapy in early NSCLC adjuvant setting as well as monotherapy in consolidation after completion of definitive chemo-radiotherapy, it has not yet been assessed in combination with radiotherapy. Anecdotal data of concurrent treatment in the palliative setting suggest acceptable safety and a good tolerability of such combination.

The NICOLAS trial was initially developed to prospectively assess the safety of checkpoint inhibition concurrently with chemo-radiotherapy.

In summary, there is a definite unmet need in multi-disciplinary care to improve the prognosis of patients diagnosed with stage III NSCLC, with a strong rationale supporting the combination of chemo-radiotherapy with anti-PD-1. A major theoretical concern is the development of pneumonitis, a rare toxicity of both radiotherapy and checkpoint inhibitors. The main aim of the ongoing current trial is therefore to evaluate the pneumonitis rate in patients being treated with chemo-radiotherapy in combination with nivolumab treatment.

Rationale for protocol amendment 2:

Since the NICOLAS trial was initiated, the landscape of combining chemo-radiotherapy with immune-checkpoint inhibition, such as anti-PD-1 antibodies, has changed rapidly, opening a new window of opportunity.

There is a very strong interest of the multidisciplinary lung cancer community to investigate the optimal integration of anti-PD-1 treatment into chemo-radiotherapy. Currently, 11 sites from 5 countries are activated for the NICOLAS trial and recruiting strongly (ahead of schedule). Using this momentum will allow us to rapidly recruit additional patients in order to reach the power to not only determine the feasibility in terms of pneumonitis grade 2 and abouve, but also to evaluate the efficacy of the concurrent treatment.

So far, during the regular safety review, the ETOP IDMC did not observe any additional toxicity compared the chemo-radiotherapy alone.

A first planned analysis of the PACIFIC trial (stage III NSCLC treated with concurrent chemotherapy and radiotherapy, followed by the anti-PD-L1 durvalumab or observation, NCT02125461) showed an increased progression-free survival (PFS), which was co-primary endpoint together with overall survival (OS). The full details are not known, yet, but it appears that the pre-clinical rationales of combined chemo-radiotherapy and anti-PD-1 treatment can be successfully transferred into clinical trials, without serious toxicities.

A recent secondary analysis of the Keynote 001 trial indicates synergistic affects of radiotherapy and immunotherapy. This international, multicentre phase I trial assessed the effect of pembrolizumab monotherapy in patients with progressive locally advanced or metastatic NSCLC. Patients were assigned to multiple expansion cohorts to allow for the inclusion of patients who were naïve to systemic therapy and those who had progression after one or two previous regimens.

The results from this study showed that the effect of pembrolizumab was significantly higher in patients who received previous radiotherapy than in patients without previous radiotherapy.

These findings were well in line with pre-clinical studies that underlined the ability of radiotherapy to enhance antitumour immune response.

In the absence of of serious pulmonary toxicity, the apperant benefit of chemo-radiotherapy and anti-PD-1 and the high interest of the NICOLAS study group, we propose to amend the NICOLAS trial protocol to expand on the number of patients in order to reach sufficient power for an efficacy readout (progression-free survival).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non small cell lung carcinoma
* Locally advanced stage IIIA or III B (T0-3 N2-3 or T4N0-3 M0) NSCLC, according to 7th TNM classification.

Within 35 days before beginning of first platinum-based chemotherapy cycle:

* Nodal status N2 or N3 must to be proven (by biopsy, EBUS, mediastinoscopy or thoracoscopy) except for overt cT4 disease.
* Whole body FDG-PET, plus contrast enhanced CT of thorax / upper Abdomen (from top of thorax until adrenal glands, and full liver and kidney included) in addition to or in combination with PET.
* Brain MRI (preferred) or high-quality brain CT with intravenous contrast at the time of staging mandatory.
* Measurable disease (according to RECIST v1.1 criteria)
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Life expectancy > 3 months
* Previous delivery of a maximum of one 3-weekly cycle of platinum-based chemotherapy
* All AEs from previous therapies (including the first chemotherapy cycle in the context of this trial) resolved to grade <2 (except fatigue, alopecia, nausea, lack of appetite and peripheral neuropathy).
* Adequate haematological function:
* WBC ≥ 2000/μL
* haemoglobin ≥ 9 g/dL
* neutrophil count ≥ 1×109/L
* platelet count ≥ 100 × 109/L
* Adequate liver function:
* Total bilirubin ≤ 1.5 x ULN (except patients with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dl)
* ALT ≤3 × ULN
* alkaline phosphatase ≤ 5 x ULN.
* Adequate renal function: Calculated creatinine clearance ≥ 30 ml/min (according to Cockroft-Gault):
* ≥60ml/min for patient receiving cisplatin
* ≥30ml/min for patient receiving carboplatin.
* Pulmonary function FEV1 of 1.0 l or > 40% predicted value and DLCO > 30% predicted value
* Patient capable of proper therapeutic compliance, and accessible to correct follow-up.
* Women of childbearing potential, including women who had their last menstrual period in the last 2 years, must have a negative serum or urine pregnancy test within 7 days before trial enrolment. The test must be repeated within 24 hours before beginning nivolumab treatment and then before every 2nd nivolumab administration. Pregnancy tests should be repeated at approximately 30 days and approximately 70 days after nivolumab treatment stops.
* Written Informed Consent (IC) for trial treatment must be signed and dated by the patient and the investigator prior to any trial-related evaluation and/or intervention.

Exclusion Criteria:

* Patient with mixed small-cell and non-small-cell histologic features
* Patient with pleural or pericardial effusions proven to be malignant
* Prior chemotherapy, radiotherapy or molecular targeted therapy for NSCLC (with the exception of one cycle of chemotherapy given prior to enrolment into this trial)
* Patients with an active, known or suspected autoimmune disease. Patients are permitted to enrol if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Patient who has had in the past 3 years any previous or concomitant malignancy EXCEPT adequately treated basal or squamous cell carcinoma of the skin, in situ carcinoma of the cervix or bladder, in situ ductal carcinoma of the breast.
* Patient with other serious diseases or clinical conditions, including but not limited to uncontrolled active infection and any other serious underlying medical processes that could affect the patient's capacity to participate in the trial.
* Ongoing clinically serious infections requiring systemic antibiotic or antiviral, antimicrobial, antifungal therapy.
* Known or suspected hypersensitivity to nivolumab or any of its excipients
* History of severe hypersensitivity reaction to any monoclonal antibody
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the trial or evaluation of the trial results.
* Established pathological diagnosis of underlying interstitial lung disease or pulmonary fibrosis
* Women who are pregnant or in the period of lactation
* Sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method during the trial treatment and for a period of at least 7 months (male participants) and 5 months (female participants) following the last administration of nivolumab.
* Patients receiving any concurrent anticancer systemic therapy
* HIV, active Hepatitis B or Hepatitis C infection
* Previous radiotherapy to the thorax (prior to inclusion), including radiotherapy for breast cancer
* Planned radiotherapy to lung of mean dose > 20 Gy or V20 > 35 %
* Patient who received treatment with an investigational drug agent during the 3 weeks before enrolment in the trial
* Metastatic disease (mandatory assessment of the brain either by MRI or high-quality CT with intravenous contrast at the time of staging as well as systemic PET and CT scan)
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-11-25 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Solange Peters, MD PhD, Study Chair — University of Lausanne Hospitals; Dirk De Ruysscher, MD PhD, Study Chair — Maastro Clinic, Maastricht, The Netherlands
Locations (11):
- University Hospital Leuven, Leuven, Belgium
- Thoracic Oncology Centre Munich, Munich, Germany
- Netherlands (2):
  - VUMC, Amsterdam
  - MAASTRO Clinic, Maastricht
- Spain (3):
  - Vall d'Hebron University Hospital, Barcelona
  - Catalan Institute of Oncology, Barcelona
  - Hospital Virgen de la Salud, Toledo
- Switzerland (4):
  - HFR Fribourg- Hôpital cantonal, Fribourg
  - Kantonsspital Winterthur, Winterthur
  - Hirslanden Klinik Zürich, Zurich
  - University Hospital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salama JK, Vokes EE. New radiotherapy and chemoradiotherapy approaches for non-small-cell lung cancer. J Clin Oncol. 2013 Mar 10;31(8):1029-38. doi: 10.1200/JCO.2012.44.5064. Epub 2013 Feb 11. PMID 23401449
- [Background] Shaverdian N, Lisberg AE, Bornazyan K, Veruttipong D, Goldman JW, Formenti SC, Garon EB, Lee P. Previous radiotherapy and the clinical activity and toxicity of pembrolizumab in the treatment of non-small-cell lung cancer: a secondary analysis of the KEYNOTE-001 phase 1 trial. Lancet Oncol. 2017 Jul;18(7):895-903. doi: 10.1016/S1470-2045(17)30380-7. Epub 2017 May 24. PMID 28551359

RESULTS

PARTICIPANT FLOW:
Groups:
- Concurrent CRT-Nivo: 4 doses of nivolumab 360mg concurrently with standard chemo-radiotherapy, followed by 480mg for up to 1 year from start of nivolumab treatment.
  Nivolumab: Nivolumab is a fully human monoclonal antibody that targets the programmed death-1 (PD-1) cell surface membrane receptor. PD-1 is a negative regulatory molecule expressed by activated T and B lymphocytes.Binding of PD-1 to its ligands, 1 (PD-L1) and 2 (PD-L2), results in the down-regulation of lymphocyte activation. Nivolumab inhibits the interaction of programmed cell death Protein 1 (PD-1)with its ligands, PD-L1 and PD-L2, resulting in enhanced T-cell proliferation.
Period: Overall Study
Arm/Group | Concurrent CRT-Nivo
Started | 79 (Only patients enrolled after protocol amendments 1 (n=43) and 2 (n=36) were analysed (concurrent CRT+Nivo). Patients who received CRT and sequentially Nivo (enrolled under original protocol (n=12) or protocol amendment 1 (n=3)) were not included in the analysis population.)
Completed | 31
Not Completed | 48
Not completed — Death (never started treatment) | 2
Not completed — Death | 2
Not completed — Progression | 20
Not completed — Adverse Event | 20
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1
Not completed — Patient did not receive treatment for more than six weeks | 1

BASELINE CHARACTERISTICS:
Arm/Group | Concurrent CRT-Nivo
Number analyzed (Participants) | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 35
Age, Continuous [Median (Full Range); unit: years] | 62 [41 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 53
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 14
  Belgium | 12
  Switzerland | 11
  Germany | 13
  Spain | 29

OUTCOME MEASURES:

1. Primary Outcome: Grade ≥3 Pneumonitis (CTCAE v4.0) up to 6 Months Post-radiotherapy
Description: It is defined as the number of patients reaching up to 6 months post-radiotherapy without any episode of CTCAE v4.0 grade ≥3 pneumonitis. It will be used as the primary endpoint for all patients followed for at least 6 months beyond radiotherapy.
Time Frame: Time from enrolment until 6 months post-radiotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Chemo-radiotherapy With Concurrent Nivolumab
Number analyzed (Participants) | 77
Participants | 71

2. Secondary Outcome: Progression-free Survival by RECIST v1.1 (PFS)
Description: PFS, κey secondary endpoint, is defined as the time from the date of enrolment until first documented progression or death, if progression is not documented. For patients without a PFS event, censoring occurs at the last tumour assessment.
  Database cutoff: 18 September 2019
Time Frame: From the date of enrolment of the first patient up to 3 years, which is also 1 year after the enrolment of the last patient (i.e., from September 2016 to September 2019)
Population: ITT cohort
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemo-radiotherapy With Concurrent Nivolumab
Number analyzed (Participants) | 79
months | 12.7 [10.1 to 22.8]

3. Secondary Outcome: (Grade ≥3) Pneumonitis-free Rate
Description: Rate of TFP3, evaluated at 1-year based on Kaplan-Meier method, where TFP3 is defined as the time from the date of enrolment until first documented pneumonitis of grade ≥3.
Time Frame: as for outcome 2
Population: Estimate of 1-year TFP3% based on the safety cohort (N=77 pts)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemo-radiotherapy With Concurrent Nivolumab
Number analyzed (Participants) | 77
percentage of participants | 87.0 [76.4 to 93.0]

4. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) is defined as the percentage of patients with objective response (OR).
  OR was determined using the Response Evaluation Criteria in Solid Tumors (RECIST v1.1). OR is defined as the best overall response (Complete Response (disappearance of all target and non-target lesions; no new lesions) or Partial Response (≥decrease in the sum of the largest diameters of target lesions; no new lesions)) across all assessment points from enrollment to termination of trial treatment. Radiological tumour assessment was performed using CT scans.
Time Frame: as for outcome 2
Population: ITT cohort
Measure: Number (95% Confidence Interval); unit: percentage of patients with OR
Arm/Group | Chemo-radiotherapy With Concurrent Nivolumab
Number analyzed (Participants) | 79
percentage of patients with OR | 73.4 [62.3 to 82.7]

5. Secondary Outcome: Time to Treatment Failure (TTF).
Description: Time to treatment failure (TTF) is defined as time from enrolment to discontinuation of trial treatment for any reason. Disease progression, treatment toxicity, death, withdrawal and lost to follow-up which occurred after treatment completion are viewed as events.
Time Frame: as for outcome 2
Population: based on ITT cohort
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemo-radiotherapy With Concurrent Nivolumab
Number analyzed (Participants) | 79
months | 9.2 [6.4 to 12.4]

6. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of enrolment until death from any cause. The patients without OS event (death) were censored at their last follow-up date
Time Frame: From the date of enrolment of the first patient up to 4 years (i.e., from September 2016 to September 2020).
Population: ITT cohort
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemo-radiotherapy With Concurrent Nivolumab
Number analyzed (Participants) | 79
months | 38.8 [26.8 to NA] — The upper 95% confidence limit is not estimable.

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from the date of first trial treatment until 100 days after the final dose of nivolumab, regardless of whether they were considered related to the trial treatment. After the last dose, only AEs considered possibly related to nivolumab had to be reported. Any known untoward event that occurred subsequent to the AE reporting period, possibly related to the protocol treatment, was considered an AE.
Description: In the 'All Cause Mortality' section, number of at risk patients includes all enrolled patients, while in the 'Serious Adverse Events' and 'Other (Not Including Serious) Adverse Events' sections, at risk patients refer to the population who received at least one dose of trial treatment.
Arm/Group | Concurrent CRT-Nivo
All-Cause Mortality (participants affected / at risk) | 37/79
Serious Adverse Events (participants affected / at risk) | 37/77
Other Adverse Events (participants affected / at risk) | 76/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concurrent CRT-Nivo (N=77)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 2 (2)
Fever (General disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Esophageal fistula (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Bronchial infection (Infections and infestations) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 13 (13)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 3 (3)
Lung infection (Infections and infestations) | 2 (2)
Stroke (Nervous system disorders) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4)
Malaise (General disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Autoimmune disorder (Immune system disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Esophageal varices hemorrhage (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Concurrent CRT-Nivo (N=77)
Anemia (Blood and lymphatic system disorders) | 36
Neutrophil count decreased (Blood and lymphatic system disorders) | 25
Vertigo (Ear and labyrinth disorders) | 4
Hypothyroidism (Endocrine disorders) | 6
Hyperthyroidism (Endocrine disorders) | 5
Dysphagia (Gastrointestinal disorders) | 26
Esophagitis (Gastrointestinal disorders) | 21
Nausea (Gastrointestinal disorders) | 17
Diarrhea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 8
Esophageal pain (Gastrointestinal disorders) | 7
Mucositis oral (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 38
Fever (General disorders) | 12
Pain (General disorders) | 12
Flu like symptoms (General disorders) | 6
Non-cardiac chest pain (General disorders) | 5
Bronchial infection (Infections and infestations) | 6
Upper respiratory infection (Infections and infestations) | 6
Lung infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 4
Dermatitis radiation (Injury, poisoning and procedural complications) | 5
Lipase increased (Investigations) | 9
Lymphocyte count decreased (Investigations) | 9
Platelet count decreased (Investigations) | 9
White blood cell decreased (Investigations) | 9
Creatinine increased (Investigations) | 8
Serum amylase increased (Investigations) | 8
Alanine aminotransferase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 5
Weight gain (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 14
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Dizziness (Nervous system disorders) | 11
Headache (Nervous system disorders) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 5
Tremor (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 13
Anxiety (Psychiatric disorders) | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 21
Productive cough (Respiratory, thoracic and mediastinal disorders) | 31
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 25
Pruritus (Skin and subcutaneous tissue disorders) | 12
Dry skin (Skin and subcutaneous tissue disorders) | 10
Rash acneiform (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-04): https://cdn.clinicaltrials.gov/large-docs/81/NCT02434081/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT02434081/SAP_001.pdf